CLINICAL TRIAL: NCT05751707
Title: The Role of HFCWO Via The Vest® Airway Clearance System in Addition to NIRT in the Treatment of Patient With Acute Respiratory Failure and Hypersecretion: Monocentric, Parallel Group, Controlled Randomized Clinical Trial
Brief Title: VICOR Study-High Frequency Chest Wall Oscillations (HFCWO) in Patients With Acute Respiratory Failure and Hypersecretion
Acronym: VICOR2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Raffaele Scala (Other)
Responsible Party: Sponsor-Investigator, Raffaele Scala, Head of Respiratory Intensive Care Unit, Ospedale San Donato
Organization: Ospedale San Donato (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICOR2
Record Dates: First submitted 2023-02-02; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Acute Respiratory Failure; Acute-on-chronic Respiratory Failure; Airway Clearance Impairment
Keywords: Acute respiratory failure; NIRT; HFCWO; Airway hypersecretion; Non Invasive Ventilation; High Flow Nasal Cannulae

STUDY DESIGN:
Intervention Model Description: Monocentric Parallel Group Controlled Randomized Clinical Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NIV+/-HFNC (non invasive ventilation +/- high flow nasal cannulae) & HFCWO (Experimental): Patient with acute or acute on chronic respiratory failure is treated with non invasive ventilation (with or without high flow nasal cannulae oxygen) AND High Frequency Chest Wall Oscillations
  Interventions: Device: High Frequency Chest Wall Oscillations via The Vest® Airway Clearance System
- NIV+/-HFNC and no HFCWO (No Intervention): Patient with acute or acute on chronic respiratory failure is treated with non invasive ventilation (with or without high flow nasal cannulae oxygen) AND NO High Frequency Chest Wall Oscillations
- HFNC & HFCWO (Experimental): Patient with acute or acute on chronic respiratory failure is treated with high flow nasal cannulae oxygen AND High Frequency Chest Wall Oscillations
  Interventions: Device: High Frequency Chest Wall Oscillations via The Vest® Airway Clearance System
- HFNC and no HFCWO (No Intervention): Patient with acute or acute on chronic respiratory failure is treated with high flow nasal cannulae oxygen AND High Frequency Chest Wall Oscillations

INTERVENTIONS:
Device: High Frequency Chest Wall Oscillations via The Vest® Airway Clearance System — High Frequency Chest Wall Oscillations via The Vest® Airway Clearance System is a clinical device which consists in a pump which generates high frequency oscillations and connected to a jacket worn by the patient, intended to facilitate airway secretions clearance by detaching them from the bronchial wall and moving them upwards in the bronchial system.
  Arms: HFNC & HFCWO; NIV+/-HFNC (non invasive ventilation +/- high flow nasal cannulae) & HFCWO

SUMMARY:
The study aims to evaluates if the treatment with HFCWO Via The Vest® Airway Clearance System, in addition to standard care in critically ill patients admitted in the Respiratory Intensive Care Unit for acute respiratory failure or acute on chronic respiratory failure and unable to manage secretions, could primarily prevent the need for bronchoscopy, and secondarily shorten duration of non invasive respiratory therapy, shorten length of stay and reduce mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute respiratory failure (ARF) or acute on chronic respiratory failure (including patients having home oxygen therapy, HFNC, NIV) both hypercapnic ARF (PaCO2 > 45 mmHg; PaO2/FiO2 <300) or hypoxaemic (PaCO2 <45 mmHg; PaO2/FiO2 <300);
* Informed consent from patient or legal tutor;
* Accessory respiratory muscles use;
* Respiratory rate above 25 apm;
* Use of non invasive respiratory therapy (NIRT) NIV+/-HFNC or HFNC alone since RICU admission
* Kelly neurological index ≤ 3
* Excessive airway mucus secretion (clinical evaluation asking the patient to cough) and inability to efficiently remove secretions (evaluated with the Cough Peak Flow (CPF) measurement. A CPF under 270 Lpm is highly suggestive of inadequate cough which prevent the patient from adequately manage and remove airway secretions.
* Cough score < 3: in the case of inability to perform CPF measurement due to poor patient collaboration, cough adequacy will be evaluated by a respiratory physiotherapy with a semiquantitative score ("Cough score") based on the measurement of sputum volume produced after coughing three times (1 point: less than 2 mL, 2 points: 2-6 mL, 3 points: more than 6 mL).

Exclusion Criteria:

* Patient unwillingness or incapability to provide informed consent
* Need for subcontinuous NIV(more than 20 hours per day)
* Kelly neurological index >3
* Cardiac arrest
* Severe haemodynamic instability (more than two amines required);
* acute coronary syndrome;
* Psychomotor agitation unresponsive to analgo-sedation (RASS> 1)
* Contraindications to HFCWO use: acute pneumothorax (even if chest drainage is not required ); severe chest wall deformities (pectus excavatum, pectus carinatum or pectus arcuatum); severe obesity (BMI >40 kg/m2); pregnancy; thoracic or abdominal surgery in the six previous weeks
* Nasal swab positivity to Sars-CoV-2
* Need for endotracheal intubation or urgent bronchoscopy for excessive airway mucus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-12-24 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Rate of patients undergoing bronchoscopy | From date of randomization until the date when the patients undergoes bronchoscopy becauase he/she is unable to spontaneously remove secretion assessed as worsening of gas exchange or of radiological appearance, whichever comes first, up to 30 days
  Bronchoscopy is required when the patient is unable to spontaneously remove secretions despite physiokinesitherapy (Cough score < 3 and gas exchange deterioration during NIRT (PaO2/FiO2<200 or PaO2 <60 and/or PaCO2 increasement of 20%) and/or radiological worsening (development of lobar/multilobar/pulmonary atelectasis or pre-existing atelectasis worsening)

SECONDARY OUTCOMES:
Days of non-invasive respiratory treatment (NIRT) duration | From date of randomization until the date when the patient no more requires NIRT because of improving gas exchange, assessed up to 30 days (days)
  Evaluates if reduction of NIRT duration in patients treated with HFCWO compared to patients treat only with NIRT, occurs
Days of RICU (respiratory intensive care unit) stay | From date of randomization until the date when the patient is clinically stable to be discharged from RICU, assessed up to 30 days (days-weeks)
  Evaluates if reduction of duration of RICU stay in patients treated with HFCWO compared to patients treat only with NIRT, occurs
Number of patients who undergo endotracheal intubation and Invasive mechanical ventilation | From date of randomization until the date when the patient intubated for acute worsening of clinical conditions, assessed during hospital stay, up to 90 days
  Evaluates if reduction of need for Invasive mechanical ventilation in patients treated with HFCWO compared to patients treat only with NIRT, occurs
Number of patients who undergo endotracheal intubation for inability to manage secretions in patients without a "do not resuscitate" (DNR) indication and RICU mortality for DNR patients | From date of randomization until the date when the patient intubated for acute worsening of clinical conditions, assessed during hospital stay, up to 90 days
Sputum volume | 10 days
Comfort in using The Vest airway clearance system in patients treated with HFCWO + NIRT | 48 hours after HFCWO treatment starting
  Likert questionnaire scale will be used to assess this outcome
Respiratory function tests 90 days after hospital discharge | 90 days after hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Donato, Arezzo, AR, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Longhini F, Bruni A, Garofalo E, Ronco C, Gusmano A, Cammarota G, Pasin L, Frigerio P, Chiumello D, Navalesi P. Chest physiotherapy improves lung aeration in hypersecretive critically ill patients: a pilot randomized physiological study. Crit Care. 2020 Aug 3;24(1):479. doi: 10.1186/s13054-020-03198-6. PMID 32746877
- [Result] Mahajan AK, Diette GB, Hatipoglu U, Bilderback A, Ridge A, Harris VW, Dalapathi V, Badlani S, Lewis S, Charbeneau JT, Naureckas ET, Krishnan JA. High frequency chest wall oscillation for asthma and chronic obstructive pulmonary disease exacerbations: a randomized sham-controlled clinical trial. Respir Res. 2011 Sep 10;12(1):120. doi: 10.1186/1465-9921-12-120. PMID 21906390
- [Result] Nicolini A, Cardini F, Landucci N, Lanata S, Ferrari-Bravo M, Barlascini C. Effectiveness of treatment with high-frequency chest wall oscillation in patients with bronchiectasis. BMC Pulm Med. 2013 Apr 4;13:21. doi: 10.1186/1471-2466-13-21. PMID 23556995
- [Result] Celik M, Yayik AM, Kerget B, Kerget F, Doymus O, Aksakal A, Ozmen S, Aslan MH, Uzun Y. High-Frequency Chest Wall Oscillation in Patients with COVID-19: A Pilot Feasibility Study. Eurasian J Med. 2022 Jun;54(2):150-156. doi: 10.5152/eurasianjmed.2022.21048. PMID 35703523
- [Result] Scala R, Naldi M, Maccari U. Early fiberoptic bronchoscopy during non-invasive ventilation in patients with decompensated chronic obstructive pulmonary disease due to community-acquired-pneumonia. Crit Care. 2010;14(2):R80. doi: 10.1186/cc8993. Epub 2010 Apr 29. PMID 20429929
- [Result] Hall GJ, Gandevia B. Relationship of the loose cough sign to daily sputum volume. Observer variation in its detection. Br J Prev Soc Med. 1971 May;25(2):109-13. doi: 10.1136/jech.25.2.109. No abstract available. PMID 5581051